CLINICAL TRIAL: NCT03255785
Title: A Prospective Evaluation of Mild to Moderate Open-Angle Glaucoma Subjects With Cataract Treated With Cataract Surgery Plus One Trabecular Micro-bypass Stent and One Suprachoroidal Stent
Brief Title: Open-Angle Glaucoma Subjects With Cataract Treated With Cataract Surgery Plus One iStent and One iStent Supra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCF-040
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: iStent and iStent Supra
Masking Description: IOP outcome masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- G1 plus G3 with phaco (Experimental): Cataract surgery via phacoemulsification followed by implantation of one iStent and one iStent Supra
  Interventions: Device: Cataract surgery plus one iStent and one iStent Supra implanted

INTERVENTIONS:
Device: Cataract surgery plus one iStent and one iStent Supra implanted — Cataract surgery via phacoemulsfication plus one iStent and one iStent supra

SUMMARY:
Open Angle Glaucoma Subjects with Cataract treated with Cataract Surgery plus one trabecular micro-bypass stent and one suprachoroidal stent

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant cataract requiring surgery Primary open-angle or pseudoexfoliative glaucoma Visual field defects no worse than -12dB Subject on two ocular hypotensive medications at screening Medicated IOP at screening between 18 and 30 mm Hg Normal iridocorneal anatomy Absence of peripheral anterior synechiae

Exclusion Criteria:

* Monocular subjects or those with wore than 20/200 vision in fellow eye Prior stent implantation, incision glaucoma surgery, or laser trabeculoplasty in study eye Traumatic, uveitic, or neovascular glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
20% IOP reduction from baseline | Month 12
  IOP measured via Goldmann tonometry in mm Hg and compared to baseline IOP

SECONDARY OUTCOMES:
IOP less than or equal to 18 mm Hg | Month 12
  IOP measured via Goldmann tonometry in mm Hg

CONTACTS AND LOCATIONS:
Locations (1):
- Glaukos Investigator Sites, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No